CLINICAL TRIAL: NCT03991377
Title: A Multicenter Phase II Rater-blinded Randomized Controlled Trial (RCT) to Compare Effectiveness of Eye Movement Desensitization Reprocessing Therapy (EMDR) vs Treatment as Usual (TAU) in First Episode Psychosis and History of Trauma.
Brief Title: A Rater-blinded RCT to Compare Effectiveness of EMDR vs TAU in Patients With First Episode Psychosis and History of Psychological Trauma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Consorci Hospitalari de Vic (Other); Hospital Mutua de Terrassa (Other); Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI18/00009
Record Dates: First submitted 2019-05-02; First posted 2019-06-19 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Psychotic Episode; Psychological Trauma
Keywords: First psychotic episode, psychological trauma, EMDR therapy, Treatment as usual
MeSH Terms: conditions — Psychological Trauma | interventions — Eye Movement Desensitization Reprocessing; Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a multicenter phase II rater-blinded randomized controlled trial with two parallel branches, EMDR + TAU and TAU, of 80 FEP patients who have a history of psychological trauma, even if they do not currently meet DSM-V criteria for PTSD.
Who Masked: Outcomes Assessor
Masking Description: Clinical raters carrying out evaluations will be blind to the participants' research condition. Patients will not be blind to treatment as a sham alternative to EMDR therapy is impossible due to its use of bilateral stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR therapy (Experimental): Patients in the psychotherapy intervention will receive up to 20 individual sessions of EMDR, weekly sessions, of 60 minutes each, using the standard EMDR therapy protocol developed by Shapiro to treat both current and past trauma-related symptom.
  Interventions: Behavioral: Eye movement desensitization and reprocessing therapy; Drug: Treatment as usual
- Treatment as usual (Active Comparator): Multidisciplinary approach that includes pharmacological treatment and psychological support.
  Interventions: Drug: Treatment as usual

INTERVENTIONS:
Behavioral: Eye movement desensitization and reprocessing therapy — EMDR is an integrative psychotherapy that uses standardized protocols and elements of cognitive-behavioral, interpersonal, and body-centered therapies, as well as dual stimulation (e.g., side-to-side eye movements).
  The current standard protocol includes eight phases:
  1. Patient history.
  2. Patient preparation.
  3. Patient assessment.
  4. Memory desensitization.
  5. Installing the positive cognition.
  6. Body scan.
  7. Closure.
  8. Reevaluation.
  Other Names: EMDR
  Arms: EMDR therapy
Drug: Treatment as usual — Once patients are discharged from hospital, they will be treated by the multidisciplinary team of the Specialized Early Intervention Programme for Incipient Psychosis (PAE-TPI) as part of their usual treatment, which consists of a multidisciplinary approach that includes pharmacological treatment and psychological support, from social workers or nursing staff. An individual care plan is drawn up depending on individual needs and may include follow-up psychiatric visits to evaluate clinical status and, if necessary, readjust pharmacological treatment, and psychological visits to assess and detect risk situations and prevent relapses using a non-trauma focused CBT. In no case will psychological treatment focus on PTSD.
  Other Names: TAU

SUMMARY:
The main objective of this project is to analyze whether EMDR therapy, as an adjuvant to usual treatment, is effective in reducing post-traumatic stress and psychotic/affective symptoms in patients with a FEP and comorbid psychological trauma associated with first hospital admission and / or previous stressful life event.

DETAILED DESCRIPTION:
Background: The experience of psychosis and hospitalization may be highly distressing. In fact, a significant proportion of FEP patients show posttraumatic stress symptoms during their recovery, which has been conceptualized as a posttraumatic postpsychotic syndrome (PPS). Moreover, the prevalence of childhood trauma in psychotic patients is four times higher than in general population. It is currently recognized the clinical implications of trauma in psychosis, as well as the need for treatment. Eye Movement Desensitization and Reprocessing (EMDR) therapy is a well stablished trauma treatment. EMDR is an eight- phase treatment protocol that includes bilateral stimulation to desensitize the discomfort caused by traumatic memories. Initial evidence suggests that EMDR is safe, well tolerated and beneficial in chronic patients with severe mental illness and comorbid psychological trauma.

Objectives: To assess if EMDR therapy leads to: 1) reduce post-traumatic stress symptoms; 2) reduce positive, negative and affective symptoms; 3) improve overall functioning; and 4) improve quality of life.

The hypothesis of this trial is that subjects of the EMDR group will experience an overall clinical improvement after therapy and will suffer from less admissions and relapses at 12 months of follow-up.

Design:

This is a multicenter phase II rater-blinded randomized controlled trial in which 80 FEP patients and psychological trauma will be randomly assigned to EMDR (n=40) or to TAU (n=40). Patients in the EMDR condition will receive up to 20 psychotherapeutic sessions of 60 minutes,

Clinical and diagnostic variables:

1. Traumatic events will be measured by Global Assessment of Posttraumatic Stress Questionnaire, Cumulative Trauma Screening, the Impact of Event Scale-Revised, the Dissociative Experiences Scale, Childhood Trauma Questionnaire, The Holmes-Rahe Life Stress Inventory and the Dissociative Experiences Questionnaire.
2. Clinical symptomatology will be assessed by using:

   * Suicide and Drug Consumption module of the International Neuropsychiatric Interview
   * Structured Clinical Interview for Positive and Negative Syndrome Scale
   * Young's Scale for Mania Evaluation
   * Beck Depression II Questionnaire.
3. Functionality will be assessed with the Global Assessment of Functioning questionnaire.
4. Cognitive insight and adherence to the treatment will be measured using the Beck Cognitive Insight Scale and the Drug Attitude Inventory.
5. Quality of Life will be assessed with the Standardized Instrument developed by the EuroQol Group.

All variables will be measured at baseline, post-treatment and 12 months of follow-up.

Randomization procedure All patients meeting the inclusion criteria will receive the baseline (T0) assessment. After T0, participants will be assigned to the EMDR or TAU group following a biased coin procedure: (1) the first two patients will be randomly allocated to EMDR with p = 0.5, (2) the next patient will be allocated as follows: (b1) if one group already includes at least two more patients than the other group, the patient will be randomly allocated to EMDR with p = 0.8 is this is the smallest group and with p = 0.2 if it is the largest group, (b2) otherwise, we will first simulate that the patient is allocated to EMDR and calculate the sum of the between-group square standardized differences in site, age, sex, diagnosis and before the clinical trial between groups, we will then simulate that the patient is allocated to TAU and recalculate the sum, and finally randomly allocate the patient to EMDR with p = 0.8 if this was associated to the smallest sum and with p = 0.2 if not. For example, if we had already included 10 patients to the EMDR group and 8 patients to the TAU group, the 19th patient would be randomly allocated with p = 0.2 for EMDR and p = 0.8 for TAU. If he/she was allocated to TAU, for the 20th patient we would calculate the above sum of covariates after simulating that the he/she is allocated to EMDR and after simulating that he/she is allocated to TAU, and if the sum of the EMDR simulation was larger than the sum of the TAU simulation, we would randomly allocate the 20th patient with p = 0.2 for EMDR and p = 0.8 for TAU. Following this procedure, the final groups should be balanced in size and matched in site, age, sex and diagnosis. All steps of the randomization process will be automatically carried out by an independent researcher in a central location using a computer program.

Computation of sample size The study aims to assess the relative efficacy of an EMDR intervention protocol for patients with PEP versus TAU mainly in stabilization and clinical improvement - reduction of anxious, depressive, somatic and/or psychotic symptoms, among others. For this reason, the main variable used is the number of clinical relapses after the intervention, with a follow-up of up to 12 months. Taking into account previous studies, the calculation of the sample size has been calculated based on a survival analysis with the statistical package "powerSurvEpi" for R, using an alpha = 0.005 instead of 0.05 to allow correction for multiple comparisons. The number of patients required to detect a hazard ratio = 2 in a Cox regression with a statistical power of 80% and alpha = 0.005 is n = 36 per intervention group (two groups, total n = 72). According to Chambless and Hollon, a sample of this size should show clinically relevant differences. Assuming a loss percentage of approximately 10-15% of the patients in the study, it would be necessary to recruit approximately 80 patients, 40 for each branch of intervention.

Statistical analysis:

In order to be able to make the relevant comparisons, it was decided to include comparisons with a control group of healthy participants in the statistical analyses.

Dropouts and follow-up:

If a participant requires an inpatient stay due to an acute episode of a psychotic disorder during the 6-month intervention period, the patient will be excluded from the trial and considered as dropout because the hospital admission will mean the patient cannot continue with the EMDR psychotherapy during the acute phase. In the case of relapse during follow-up, patients will be maintained in the trial to obtain maximum information on the course of the illness.

ELIGIBILITY:
Inclusion Criteria:

* age ≥16 years old
* presence of one or more traumatic events, causing symptoms associated with the trauma (Impact of Event Scale-Revised >0 and Subjective Units of Distress >5), but it is not necessary that traumatic events meet DSM-5 criteria for PTSD
* psychotic symptoms/psychiatric hospitalization will be considered a traumatic event when the criteria for a trauma-related disorder or stress factors according to DSM-V (Post-Traumatic Stress Disorder, Acute Stress Disorder, and Other Trauma-related Disorder and unspecified stress factors) are also met
* ability to read and write in Spanish.

Exclusion Criteria:

* current suicidal risk
* presence of organic brain diseases
* have received trauma-focused therapy in the past 2 years.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of the severity of trauma-related symptoms | Change from baseline to visits at 6 and 12 months
  To measure severity and changes in trauma-related symptoms with the Impact of Event Scale - Revised. Items are rated on a 5-point Likert scale ranging from 0 and 4, yielding a total score ranging from 0 to 88.

SECONDARY OUTCOMES:
Making a PTSD diagnosis | Change from baseline to visits at 6 and 12 months
  To diagnose PTSD with the Global Assessment of Posttraumatic Stress Questionnaire. Higher scores indicate more severity in trauma-related symptoms.
Detection of dissociative symptoms | Change from baseline to visits at 6 and 12 months
  To assess dissociative symptoms with the Dissociative Experiences Scale. An overall mean score ranging from 0 to 100. The higher score, the higher the severity of the dissociative symptoms.
Detection of Childhood life traumatic events | Childhood period. It is administered only during the baseline visit.
  To assess life events with the Childhood Trauma Questionnaire. A 5-point Likert scale is used, ranging from "Never True" to "Very Often True".
Detection of traumatic events in the last year | The last year. It is administered only during the baseline visit.
  To assess events with The Holmes-Rahe Life Stress Inventory. Scores below 150 reflect low levels of stress, scores between 150 and 299 represent a 50% risk of a stress-related illness in the near future and scores above 300 represent an 80% risk.
Reduction of positive psychotic symptoms | Change from baseline to visits at 6 and 12 months
  To measure changes in the Positive and Negative Syndrome Scale (PANSS) . It ranges from 7 to 49: the higher the score, the worse the positive psychotic symptoms.
Reduction in depressive symptoms | Change from baseline to visits at 6 and 12 months
  To measure changes in the Beck Depression II Questionnaire. Total scores range from 0 to 52: the higher the score, the worse the depressive symptoms.
Reduction of (hypo) manic symptoms | Change from baseline to visits at 6 and 12 months
  To measure changes in the Young Mania Rating Scale. It ranges from 0 to 130: the higher the score, the worse the manic symptoms.
Improvement of global functioning | Change from baseline to visits at 6 and 12 months
  To measure changes with the Global Assessment of Functioning Scale. The global score ranges from 0 to 100. The higher the score, the higher the functional status.
Improving of the quality of life associated with health | Change from baseline to visits at 6 and 12 months
  To measure changes with the Standardized Instrument for Evaluating Quality of Life Associated with Health.The global score ranging from 0 to 100. The lower scores indicate poorer awareness of the quality of life associated with health.
Improving awareness of having a mental disorder and of their need for treatment | Change from baseline to visits at 6 and 12 months
  To measure changes in the with the Beck Cognitive Insight Scale. The total score ranging from 0 to 45. The higher score on the scale, the lower severity of negative symptomatology.
Improving adherence to pharmacological treatment | Change from baseline to visits at 6 and 12 months
  To measure changes in the attitude towards medication with the Drug Attitude Inventory. The total score can oscillate between 10 and 20. The higher the score, the more positive the perceived effect of the medication.
Reducing in the number of relapses | Change from baseline to visits at 6 and 12 months
  To measure relapses with the register of the number hospital admissions and/or emergency visits

CONTACTS AND LOCATIONS:
Overall Officials: BENEDIKT L AMANN, PhD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Parc de Salut Mar, Barcelona, Spain

REFERENCES:
- [Background] Abdel-Baki A, Ouellet-Plamondon C, Malla A. Pharmacotherapy challenges in patients with first-episode psychosis. J Affect Disord. 2012;138 Suppl:S3-14. doi: 10.1016/j.jad.2012.02.029. Epub 2012 Mar 9. PMID 22405590
- [Background] Abdelghaffar W, Ouali U, Jomli R, Zgueb Y, Nacef F. Posttraumatic Stress Disorder in First-Episode Psychosis: Prevalence and Related Factors. Clin Schizophr Relat Psychoses. 2018 Fall;12(3):105-112B. Epub 2016 Jan 18. PMID 26780602
- [Background] Alvarez MJ, Roura P, Oses A, Foguet Q, Sola J, Arrufat FX. Prevalence and clinical impact of childhood trauma in patients with severe mental disorders. J Nerv Ment Dis. 2011 Mar;199(3):156-61. doi: 10.1097/NMD.0b013e31820c751c. PMID 21346485
- [Background] Báguena, M., Villarroya, E., Beleña, Á., Díaz, A., Roldán, C., and Reig, R. (2001). Propiedades Psycometricas de la Version Española de la Escala Revisionada de Impacto del Estresor (EIE-R). Anal. y Modif. Conduct. 27, 581-604.
- [Background] Bailey T, Alvarez-Jimenez M, Garcia-Sanchez AM, Hulbert C, Barlow E, Bendall S. Childhood Trauma Is Associated With Severity of Hallucinations and Delusions in Psychotic Disorders: A Systematic Review and Meta-Analysis. Schizophr Bull. 2018 Aug 20;44(5):1111-1122. doi: 10.1093/schbul/sbx161. PMID 29301025
- [Background] Beattie N, Shannon C, Kavanagh M, Mulholland C. Predictors of PTSD symptoms in response to psychosis and psychiatric admission. J Nerv Ment Dis. 2009 Jan;197(1):56-60. doi: 10.1097/NMD.0b013e31819273a8. PMID 19155811
- [Background] Beck AT, Baruch E, Balter JM, Steer RA, Warman DM. A new instrument for measuring insight: the Beck Cognitive Insight Scale. Schizophr Res. 2004 Jun 1;68(2-3):319-29. doi: 10.1016/S0920-9964(03)00189-0. PMID 15099613
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Bendall S, Alvarez-Jimenez M, Hulbert CA, McGorry PD, Jackson HJ. Childhood trauma increases the risk of post-traumatic stress disorder in response to first-episode psychosis. Aust N Z J Psychiatry. 2012 Jan;46(1):35-9. doi: 10.1177/0004867411430877. PMID 22247091
- [Background] Bernstein DP, Fink L, Handelsman L, Foote J, Lovejoy M, Wenzel K, Sapareto E, Ruggiero J. Initial reliability and validity of a new retrospective measure of child abuse and neglect. Am J Psychiatry. 1994 Aug;151(8):1132-6. doi: 10.1176/ajp.151.8.1132. PMID 8037246
- [Background] Bernstein EM, Putnam FW. Development, reliability, and validity of a dissociation scale. J Nerv Ment Dis. 1986 Dec;174(12):727-35. doi: 10.1097/00005053-198612000-00004. PMID 3783140
- [Background] Berry K, Ford S, Jellicoe-Jones L, Haddock G. Trauma in relation to psychosis and hospital experiences: the role of past trauma and attachment. Psychol Psychother. 2015 Sep;88(3):227-39. doi: 10.1111/papt.12035. Epub 2014 Jul 15. PMID 25044987
- [Background] Bobes., J. (1998). A Spanish validation study of the MINI International Neuropsychiatric Interview. SEC55.Diagnostic tools Prim. care psychiatry, 198s-199s.
- [Background] Chambless DL, Hollon SD. Defining empirically supported therapies. J Consult Clin Psychol. 1998 Feb;66(1):7-18. doi: 10.1037//0022-006x.66.1.7. PMID 9489259
- [Background] Colom F, Vieta E, Martinez-Aran A, Garcia-Garcia M, Reinares M, Torrent C, Goikolea JM, Banus S, Salamero M. [Spanish version of a scale for the assessment of mania: validity and reliability of the Young Mania Rating Scale]. Med Clin (Barc). 2002 Sep 28;119(10):366-71. doi: 10.1016/s0025-7753(02)73419-2. Spanish. PMID 12372167
- [Background] Fusar-Poli P, McGorry PD, Kane JM. Improving outcomes of first-episode psychosis: an overview. World Psychiatry. 2017 Oct;16(3):251-265. doi: 10.1002/wps.20446. PMID 28941089
- [Background] Gibson LE, Alloy LB, Ellman LM. Trauma and the psychosis spectrum: A review of symptom specificity and explanatory mechanisms. Clin Psychol Rev. 2016 Nov;49:92-105. doi: 10.1016/j.cpr.2016.08.003. Epub 2016 Aug 31. PMID 27632064
- [Background] Gonzalez-Vazquez AI, Del Rio-Casanova L, Seijo-Ameneiros N, Cabaleiro-Fernandez P, Seoane-Pillado T, Justo-Alonso A, Santed-German MA. Validity and reliability of the Spanish version of the Somatoform Dissociation Questionnaire (SDQ-20). Psicothema. 2017 May;29(2):275-280. doi: 10.7334/psicothema2016.346. PMID 28438254
- [Background] González de Rivera, J. L., and Morera Fumero, A. (1983). La valoración de sucesos vitales : Adaptación española de la escala de Holmes y Rahe. Psiquis (Mexico). 4, 7-11.
- [Background] Gutierrez-Zotes JA, Valero J, Cortes MJ, Labad A, Ochoa S, Ahuir M, Carlson J, Bernardo M, Canizares S, Escartin G, Canete J, Gallo P, Salamero M. Spanish adaptation of the Beck Cognitive Insight Scale (BCIS) for schizophrenia. Actas Esp Psiquiatr. 2012 Jan-Feb;40(1):2-9. Epub 2012 Jan 1. PMID 22344490
- [Background] Hall RC. Global assessment of functioning. A modified scale. Psychosomatics. 1995 May-Jun;36(3):267-75. doi: 10.1016/S0033-3182(95)71666-8. PMID 7638314
- [Background] Hernandez A, Gallardo-Pujol D, Pereda N, Arntz A, Bernstein DP, Gaviria AM, Labad A, Valero J, Gutierrez-Zotes JA. Initial validation of the Spanish childhood trauma questionnaire-short form: factor structure, reliability and association with parenting. J Interpers Violence. 2013 May;28(7):1498-518. doi: 10.1177/0886260512468240. Epub 2012 Dec 24. PMID 23266990
- [Background] Hernandez G, Garin O, Pardo Y, Vilagut G, Pont A, Suarez M, Neira M, Rajmil L, Gorostiza I, Ramallo-Farina Y, Cabases J, Alonso J, Ferrer M. Validity of the EQ-5D-5L and reference norms for the Spanish population. Qual Life Res. 2018 Sep;27(9):2337-2348. doi: 10.1007/s11136-018-1877-5. Epub 2018 May 16. PMID 29767329
- [Background] Hogan TP, Awad AG, Eastwood R. A self-report scale predictive of drug compliance in schizophrenics: reliability and discriminative validity. Psychol Med. 1983 Feb;13(1):177-83. doi: 10.1017/s0033291700050182. PMID 6133297
- [Background] Holmes TH, Rahe RH. The Social Readjustment Rating Scale. J Psychosom Res. 1967 Aug;11(2):213-8. doi: 10.1016/0022-3999(67)90010-4. No abstract available. PMID 6059863
- [Background] http://www.who.int/mediacentre/news/releases/2013/trauma_mental_health_20130806/es/ (2013).
- [Background] https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/ (2019).
- [Background] Icaran E, Colom R, Orengo-Garcia F. [Validation study of the dissociative experiences scale in Spanish population sample]. Actas Luso Esp Neurol Psiquiatr Cienc Afines. 1996 Jan-Feb;24(1):7-10. Spanish. PMID 8900971
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Lecomte T, Spidel A, Leclerc C, MacEwan GW, Greaves C, Bentall RP. Predictors and profiles of treatment non-adherence and engagement in services problems in early psychosis. Schizophr Res. 2008 Jul;102(1-3):295-302. doi: 10.1016/j.schres.2008.01.024. Epub 2008 Mar 4. PMID 18295458
- [Background] Lingjaerde O, Ahlfors UG, Bech P, Dencker SJ, Elgen K. The UKU side effect rating scale. A new comprehensive rating scale for psychotropic drugs and a cross-sectional study of side effects in neuroleptic-treated patients. Acta Psychiatr Scand Suppl. 1987;334:1-100. doi: 10.1111/j.1600-0447.1987.tb10566.x. No abstract available. PMID 2887090
- [Background] María Crespo y Ma Mar Gómez (2012). Posttraumatic Stress Assessment: Introducing the Global Assessment of Posttraumatic Stress Questionnaire. Clínica y Salud 23, 25-41.
- [Background] McEvoy JP, Freter S, Everett G, Geller JL, Appelbaum P, Apperson LJ, Roth L. Insight and the clinical outcome of schizophrenic patients. J Nerv Ment Dis. 1989 Jan;177(1):48-51. doi: 10.1097/00005053-198901000-00008. PMID 2535871
- [Background] McGorry PD, Chanen A, McCarthy E, Van Riel R, McKenzie D, Singh BS. Posttraumatic stress disorder following recent-onset psychosis. An unrecognized postpsychotic syndrome. J Nerv Ment Dis. 1991 May;179(5):253-8. doi: 10.1097/00005053-199105000-00002. PMID 1781819
- [Background] McGrath JJ, Saha S, Lim CCW, Aguilar-Gaxiola S, Alonso J, Andrade LH, Bromet EJ, Bruffaerts R, Caldas de Almeida JM, Cardoso G, de Girolamo G, Fayyad J, Florescu S, Gureje O, Haro JM, Kawakami N, Koenen KC, Kovess-Masfety V, Lee S, Lepine JP, McLaughlin KA, Medina-Mora ME, Navarro-Mateu F, Ojagbemi A, Posada-Villa J, Sampson N, Scott KM, Tachimori H, Ten Have M, Kendler KS, Kessler RC; WHO World Mental Health Survey Collaborators. Trauma and psychotic experiences: transnational data from the World Mental Health Survey. Br J Psychiatry. 2017 Dec;211(6):373-380. doi: 10.1192/bjp.bp.117.205955. Epub 2017 Nov 2. PMID 29097400
- [Background] Nielsen RE, Lindstrom E, Nielsen J, Levander S. DAI-10 is as good as DAI-30 in schizophrenia. Eur Neuropsychopharmacol. 2012 Oct;22(10):747-50. doi: 10.1016/j.euroneuro.2012.02.008. Epub 2012 Mar 21. PMID 22440974
- [Background] Nijenhuis ER, Spinhoven P, Van Dyck R, Van der Hart O, Vanderlinden J. The development and psychometric characteristics of the Somatoform Dissociation Questionnaire (SDQ-20). J Nerv Ment Dis. 1996 Nov;184(11):688-94. doi: 10.1097/00005053-199611000-00006. PMID 8955682
- [Background] Novo P, Landin-Romero R, Radua J, Vicens V, Fernandez I, Garcia F, Pomarol-Clotet E, McKenna PJ, Shapiro F, Amann BL. Eye movement desensitization and reprocessing therapy in subsyndromal bipolar patients with a history of traumatic events: a randomized, controlled pilot-study. Psychiatry Res. 2014 Sep 30;219(1):122-8. doi: 10.1016/j.psychres.2014.05.012. Epub 2014 May 15. PMID 24880581
- [Background] Peralta Martin V, Cuesta Zorita MJ. [Validation of positive and negative symptom scale (PANSS) in a sample of Spanish schizophrenic patients]. Actas Luso Esp Neurol Psiquiatr Cienc Afines. 1994 Jul-Aug;22(4):171-7. Spanish. PMID 7810373
- [Background] Robles Garcia R, Salazar Alvarado V, Paez Agraz F, Ramirez Barreto F. [Assessment of drug attitudes in patients with schizophrenia: psychometric properties of the DAI Spanish version]. Actas Esp Psiquiatr. 2004 May-Jun;32(3):138-42. Spanish. PMID 15168263
- [Background] Roche E, Madigan K, Lyne JP, Feeney L, O'Donoghue B. The therapeutic relationship after psychiatric admission. J Nerv Ment Dis. 2014 Mar;202(3):186-92. doi: 10.1097/NMD.0000000000000102. PMID 24566503
- [Background] Ronconi JM, Shiner B, Watts BV. Inclusion and exclusion criteria in randomized controlled trials of psychotherapy for PTSD. J Psychiatr Pract. 2014 Jan;20(1):25-37. doi: 10.1097/01.pra.0000442936.23457.5b. PMID 24419308
- [Background] Sajatovic M, Gaur R, Tatsuoka C, De Santi S, Lee N, Laredo J, Tripathi S. Rater Training for a Multi-Site, International Clinical Trial: What Mood Symptoms may be most Difficult to Rate? Psychopharmacol Bull. 2011 Sep 15;44(3):5-14. doi: 10.64719/pb.4074. PMID 27738359
- [Background] Shapiro, F. (2001). Eye movement desensitization and reprocessing: Basic principles, protocols, and procedures (2nd ed.). Available at: http://proxy.library.nd.edu/login?url=http://search.proquest.com/docview/619595584?accountid=12874 LA - English.
- [Background] Shapiro F, Maxfield L. Eye Movement Desensitization and Reprocessing (EMDR): information processing in the treatment of trauma. J Clin Psychol. 2002 Aug;58(8):933-46. doi: 10.1002/jclp.10068. PMID 12115716
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Spidel A, Lecomte T, Kealy D, Daigneault I. Acceptance and commitment therapy for psychosis and trauma: Improvement in psychiatric symptoms, emotion regulation, and treatment compliance following a brief group intervention. Psychol Psychother. 2018 Jun;91(2):248-261. doi: 10.1111/papt.12159. Epub 2017 Oct 4. PMID 28976056
- [Background] Tarrier N, Khan S, Cater J, Picken A. The subjective consequences of suffering a first episode psychosis: trauma and suicide behaviour. Soc Psychiatry Psychiatr Epidemiol. 2007 Jan;42(1):29-35. doi: 10.1007/s00127-006-0127-2. Epub 2006 Nov 2. PMID 17082897
- [Background] Valiente-Gomez A, Moreno-Alcazar A, Treen D, Cedron C, Colom F, Perez V, Amann BL. EMDR beyond PTSD: A Systematic Literature Review. Front Psychol. 2017 Sep 26;8:1668. doi: 10.3389/fpsyg.2017.01668. eCollection 2017. PMID 29018388
- [Background] van den Berg DP, de Bont PA, van der Vleugel BM, de Roos C, de Jongh A, van Minnen A, van der Gaag M. Trauma-Focused Treatment in PTSD Patients With Psychosis: Symptom Exacerbation, Adverse Events, and Revictimization. Schizophr Bull. 2016 May;42(3):693-702. doi: 10.1093/schbul/sbv172. Epub 2015 Nov 24. PMID 26609122
- [Background] van den Berg DP, van der Gaag M. Treating trauma in psychosis with EMDR: a pilot study. J Behav Ther Exp Psychiatry. 2012 Mar;43(1):664-71. doi: 10.1016/j.jbtep.2011.09.011. Epub 2011 Sep 17. PMID 21963888
- [Background] van den Berg DP, de Bont PA, van der Vleugel BM, de Roos C, de Jongh A, Van Minnen A, van der Gaag M. Prolonged exposure vs eye movement desensitization and reprocessing vs waiting list for posttraumatic stress disorder in patients with a psychotic disorder: a randomized clinical trial. JAMA Psychiatry. 2015 Mar;72(3):259-67. doi: 10.1001/jamapsychiatry.2014.2637. PMID 25607833
- [Background] Varese F, Smeets F, Drukker M, Lieverse R, Lataster T, Viechtbauer W, Read J, van Os J, Bentall RP. Childhood adversities increase the risk of psychosis: a meta-analysis of patient-control, prospective- and cross-sectional cohort studies. Schizophr Bull. 2012 Jun;38(4):661-71. doi: 10.1093/schbul/sbs050. Epub 2012 Mar 29. PMID 22461484
- [Background] Vázquez, C., and Sanz, J. (1999). Fiabilidad y validez de la versión española del Inventario para la Depresión de Beck de 1978 en pacientes con trastornos psicológicos. Clínica y Salud 10, 59-81.
- [Background] Weber K, Giannakopoulos P, Herrmann FR, Bartolomei J, Digiorgio S, Ortiz Chicherio N, Delaloye C, Ghisletta P, Lecerf T, De Ribaupierre A, Canuto A. Stressful life events and neuroticism as predictors of late-life versus early-life depression. Psychogeriatrics. 2013 Dec;13(4):221-8. doi: 10.1111/psyg.12024. Epub 2013 Oct 28. PMID 24289463
- [Background] Weiss, D. S., and Marmar, C. R. (1997a). The Impact of Event Scale-Revised. doi:10.1007/978-0-387-70990-1_10.
- [Background] Weiss, D. S., and Marmar, C. R. (1997b). "The Impact of Event Scale-Revised.," in Assessing psychological trauma and PTSD, 399-411.
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry. 1978 Nov;133:429-35. doi: 10.1192/bjp.133.5.429. PMID 728692
- [Derived] Valiente-Gomez A, Pujol N, Moreno-Alcazar A, Radua J, Monteagudo-Gimeno E, Gardoki-Souto I, Hogg B, Alvarez MJ, Safont G, Lupo W, Perez V, Amann BL; FEP-EMDR Research Group. A Multicenter Phase II RCT to Compare the Effectiveness of EMDR Versus TAU in Patients With a First-Episode Psychosis and Psychological Trauma: A Protocol Design. Front Psychiatry. 2020 Feb 5;10:1023. doi: 10.3389/fpsyt.2019.01023. eCollection 2019. PMID 32116827